CLINICAL TRIAL: NCT00142363
Title: The DNA and Cell Bank of IFR of Neurosciences: Clinical and Genetic Study of Parkinson's Disease and Epilepsies
Brief Title: Cohorts and Collections: Clinical and Genetic Study of Parkinson's Disease and Epilepsies
Status: Terminated | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Ministry of Health, France (Other Government)
Other Study IDs: 4CH03G
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2006-03-01 (Estimated); Status verified 2006-02

CONDITIONS: Parkinson's Disease; Epilepsy
Keywords: Parkinson's disease; Parkin; Epilepsy; Phenotype-genotype correlations; Ionic channels
MeSH Terms: conditions — Parkinson Disease; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The DNA and Cell Bank of Instituts Federatifs de Recherche (IFR) of Neurosciences has been running for the last 15 years at the Institut National de la Santé Et de la Recherche Médicale (INSERM) Unit 679 (former unit 289). Since its creation, this structure has been the support of research projects in genetics for neurological and psychiatric disorders. The cohorts established have led to discoveries in monogenic disorders, such as cerebellar ataxias, spastic paraplegias, frontotemporal dementias, epilepsies, Parkinson's and Alzheimer's disease, Charcot-Marie-Tooth disease and related entities. The research projects based on the study of the genetic bases in Parkinson's disease and epilepsies are especially developed for this grant.

Concerning Parkinson's disease, the project is based on the extension of the existing cohort throughout the French Parkinson's Disease Study Group network. Concerning epilepsies, this project is the occasion to build this network with the constitution of a new cohort.

The specific aims of the scientific projects are the following for Parkinson's disease:

* to evaluate the frequency, the nature and the phenotype associated with parkin mutations in familial or sporadic forms of the disease, according to the age at onset, and
* to identify the genetic susceptibility factors in Parkinson's disease with the study of affected sibpairs and with case/controls association studies.

For epilepsies, the aims are:

* to evaluate the frequency, the nature and the phenotype associated with SCN1A, SCNab and GABR2 gene mutations in familial or sporadic forms of the affection associated with febrile seizures, and
* to search for an intervention SCN1A, SCN1B and GABRG2 as susceptible genes in these forms of epilepsies.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with Parkinson's disease, with a family history or not,
* Minors presenting clinical signs of the disease,
* Controls (without signs of the disease), matched by sex and age with the patients,
* Relatives for the familial cases,
* Patients presenting with an epilepsy episode (myoclonic epilepsy of the newborn, with febrile seizures, of the frontal lobe)

Exclusion Criteria:

* Lack of signed informed consent

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1700
Dates: Start 2004-05; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Brice, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, University Paris 6
Locations (15):
- France (15):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Hôpital Roger Salengro, Lille
  - Hôpital Neurologique Pierre Wertheimer, Lyon
  - Hôpital René et Guillaume Laennec, Nantes
  - Hôpital Pasteur, Nice
  - Hôpital Saint-Antoine, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Pitié-Salpêtrière Hospital - Centre of Clinical Investigations, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Hôpital Pontchaillou, Rennes
  - Hôpital Civil, Strasbourg
  - Hôpital Purpan, Toulouse

REFERENCES:
- [Result] Ibanez P, Bonnet AM, Debarges B, Lohmann E, Tison F, Pollak P, Agid Y, Durr A, Brice A. Causal relation between alpha-synuclein gene duplication and familial Parkinson's disease. Lancet. 2004 Sep 25-Oct 1;364(9440):1169-71. doi: 10.1016/S0140-6736(04)17104-3. PMID 15451225
- [Result] Lesage S, Leutenegger AL, Ibanez P, Janin S, Lohmann E, Durr A, Brice A; French Parkinson's Disease Genetics Study Group. LRRK2 haplotype analyses in European and North African families with Parkinson disease: a common founder for the G2019S mutation dating from the 13th century. Am J Hum Genet. 2005 Aug;77(2):330-2. doi: 10.1086/432422. No abstract available. PMID 16145815
- [Result] Lesage S, Ibanez P, Lohmann E, Pollak P, Tison F, Tazir M, Leutenegger AL, Guimaraes J, Bonnet AM, Agid Y, Durr A, Brice A; French Parkinson's Disease Genetics Study Group. G2019S LRRK2 mutation in French and North African families with Parkinson's disease. Ann Neurol. 2005 Nov;58(5):784-7. doi: 10.1002/ana.20636. PMID 16240353
- [Result] Lesage S, Leutenegger AL, Brice A. [LRRK2: a gene belonging to the ROCO family is implicated in the Parkinson's disease]. Med Sci (Paris). 2005 Dec;21(12):1015-7. doi: 10.1051/medsci/200521121015. No abstract available. French. PMID 16324633
- [Result] Ibanez P, Lesage S, Lohmann E, Thobois S, De Michele G, Borg M, Agid Y, Durr A, Brice A; French Parkinson's Disease Genetics Study Group. Mutational analysis of the PINK1 gene in early-onset parkinsonism in Europe and North Africa. Brain. 2006 Mar;129(Pt 3):686-94. doi: 10.1093/brain/awl005. Epub 2006 Jan 9. PMID 16401616
- [Result] Lesage S, Durr A, Tazir M, Lohmann E, Leutenegger AL, Janin S, Pollak P, Brice A; French Parkinson's Disease Genetics Study Group. LRRK2 G2019S as a cause of Parkinson's disease in North African Arabs. N Engl J Med. 2006 Jan 26;354(4):422-3. doi: 10.1056/NEJMc055540. No abstract available. PMID 16436781
- See also: Related Info — http://www.inserm.fr